CLINICAL TRIAL: NCT05186545
Title: An Exploratory Study of Surufatinib Combined With Chidamide and Fulvestrant in HR Positive Unresectable Metastatic Breast Cancer Refractory to Endocrine Therapy
Brief Title: An Exploratory Study of Surufatinib Combined With Chidamide and Fulvestrant in HR Positive Unresectable Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hong Zong, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-R101
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Breast Cancer Female
MeSH Terms: conditions — Breast Neoplasms | interventions — surufatinib; Fulvestrant; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): surufatinib + fulvestrant + chidamide
  Interventions: Drug: surufatinib + fulvestrant + chidamide

INTERVENTIONS:
Drug: surufatinib + fulvestrant + chidamide — surufatinib: 250 mg/d, QD PO; Fulvestrant: 500mg, im, Q4W; Chidamide 30mg, PO, BIW; Q4W

SUMMARY:
This is a prospective, single center, single arm phase II study designed to explore the efficacy and safety of surufatinib + fulvastrant + chidamide combinational treatment in HR positive breast cancer refractory to endocrine therapy.

DETAILED DESCRIPTION:
This is a prospective, single center, single arm phase II study. In the safety lead-in stage, 6 subjects will be recruited and administered with surufatinib 250 mg/d, QD PO; Fulvestrant 500mg, im, Q4W; Chidamide 30mg, PO, BIW, with four weeks as a cycle. DLTs of the 6 subjects will be evaluated in the first cycle to determine the recommended dosage of combinational therapy. Then 57 subjects will be recruited and administered with the triplet regimen to explore the efficacy and safety of combinational treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form;
* 18-75 Years (concluding 18 and 75 Years), female;
* Pathologically and cytologically confirmed non-resectable stage IV Her2 negative, HR positive (ER+ and / or PR+) breast cancer;
* Relapsed or progressed after at least first-line endocrine therapy, with patients of primary endocrine resistance excluded (patients of recurrence and metastasis progressed more than 6 months after receiving endocrine therapy or more than 2 years after receiving adjuvant endocrine therapy are eligible; patients progressed more than 1 year but less than 2 years after adjuvant endocrine therapy are not eligible);
* 2 weeks or more from the last endocrine therapy and 3 weeks or more from the last chemotherapy before enrollment;
* At least one measurable lesion is required;
* Life expectancy greater than 3 months;
* ECOG(Eastern Cooperative Oncology Group): 0~1;
* Sufficient organ and bone marrow functions as follows:

Absolute Neutrophil Count (ANC) ≥1.5×10^9/L; Platelet Count of ≥100×10^9/L; Hemoglobin≥90g/L; Total Bilirubin (TBIL)<1.5 x ULN; ALT and AST<1.5 x ULN; Serum Creatinine (SCr)<1.5×ULN; Endogenous creatinine clearance rate ≥50ml / min (Cockcroft Gault formula)

Exclusion Criteria:

* Previous treatment with VEGFR inhibitor, HDAC inhibitor or fulvestrant;
* Organ surgery performed 6 weeks before enrollment;
* A history of other malignancies within 5 years prior to enrollment, except for cervical carcinoma in situ, basal or squamous cell skin cancer;
* Known hypersensitivity to any of the study drugs or excipients;
* Hypertension that is not controlled by the drug, and is defined as: SBP ≥150 mmHg and/or DBP ≥90 mmHg;
* International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN;
* Poorly controlled diabetes before enrollment;
* Clinically significant electrolyte abnormalities judged by researchers;
* With any diseases or conditions that affected drug absorption, or the patient could not take drugs orally;
* Patients with obvious evidence of bleeding tendency or medical history or hemoptysis within 3 months before enrollment, thromboembolism within 12 months;
* Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%;
* Active infection or serious infection that is not controlled by drug (≥CTCAE v5.0 Grade 2）;
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×10^4/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×10^3/m);
* Women who are pregnant or lactating;
* Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0g;
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions, which according to the judgment of the investigator, it is reasonable to suspect that the patient is not suitable for the use of the study drug.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
ORR | up to 3 years
  The proportion of patients with a confirmed complete response or partial response on two consecutive occasions≥4 weeks apart.
DCR | up to 3 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD).
OS | up to 3 years
  The time from recruitment to death due to any cause.
Adverse Events (AEs) | up to 3 years
  Adverse events (AEs) categorized by severity in accordance with the NCI CTC AE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anyang Tumor Hospital, Anyang
  - Henan University of Science and Technology First Affiliated Hospital, Luoyang
  - Nanyang Second General Hospital, Nanyang
  - He'nan Cancer Hospital, Zhengzhou
  - The Third People's Hospital of Zhengzhou, Zhengzhou